CLINICAL TRIAL: NCT04824937
Title: A Phase II Study of the Glutaminase Inhibitor Telaglenastat (CB-839) in Combination With the PARP Inhibitor Talazoparib in Participants With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Telaglenastat + Talazoparib In Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Calithera Biosciences, Inc (Industry); Pfizer (Industry); Prostate Cancer Foundation (Other)
Responsible Party: Principal Investigator, Richard J. Lee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-325
Record Dates: First submitted 2021-02-08; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer Metastatic
Keywords: Prostate Cancer Metastatic
MeSH Terms: interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telaglenastat + Talazoparib (Experimental): During 28 day study cycles, participants will receive:
  * Telaglenastat 2x daily at a predetermined dose
  * Talazoparib 1x daily at a predetermined dose
  Interventions: Drug: Telaglenastat; Drug: Talazoparib
- Telaglenastat + Talazoparib Staggered (Experimental): If a beneficial response is seen with the Arm 1 Telaglenastat + Talazoparib combination, participants will receive telaglenastat alone 2x daily at a predetermined dose with the addition of talazoparib at 1x daily at a predetermined dose if the disease gets worse.
  Interventions: Drug: Telaglenastat; Drug: Talazoparib

INTERVENTIONS:
Drug: Telaglenastat — Capsule, taken by mouth
  Other Names: CB 839
Drug: Talazoparib — Capsule, taken by mouth
  Other Names: Taken orally

SUMMARY:
The purpose of this research is to test the effectiveness of an experimental drug combination for people with metastatic castration-resistant prostate cancer (mCRPC).

The names of the study drugs involved in this study are:

* Telaglenastat (CB-839)
* Talazoparib

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial, researching the effectiveness of the combination of telaglenastat and talazoparib in participants with metastatic castration-resistant prostate cancer (mCRPC).

The U.S. Food and Drug Administration (FDA) has not approved telaglenastat or the combination of telaglenastat and talazoparib as a treatment for any disease.

The FDA has not approved talazoparib for metastatic castration-resistant prostate cancer (mCRPC) but it has been approved for other uses.

Telaglenastat is a drug designed to stop cancer growth by blocking glutaminase activity. Glutaminase is an enzyme in the body that is overproduced by some cancers and can fuel cancer growth. Telaglenastat can lower or block glutaminase and may slow the growth or spread of some cancers.

Talazoparib is a drug that interferes with the repair activity of proteins called poly adenosine diphosphate ribose polymerases (PARP), which are found in normal and cancer cells and are involved in the repair of DNA - the genetic material found in every cell. This interference may lead to increased amounts of DNA defects and cancer cell death which may help to slow the growth of cancer cells.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

There are different points in this study in which participation will start. The first group of participants will receive the combination of telaglenastat and talazoparib for the entirety of the study. If telaglenastat plus talazoparib is beneficial to the first group this will lead to the enrollment of the next group, since telaglenastat as a single drug has not been evaluated in prostate cancer. The next group will receive telaglenastat alone with the addition of talazoparib if the disease gets worse.

It is expected that about 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed diagnosis adenocarcinoma of the prostate.
* Prostate cancer must be metastatic as confirmed by CT, PET scan, and/or bone scan.
* Prior biopsy of metastatic lesion (bone, lymph node, or visceral metastasis) with sufficient tissue for molecular analysis, or consent for a fresh biopsy for molecular analysis
* Participants must have tested negative for homologous recombination (HR) mutations (including known deleterious mutations in BRCA1, BRCA2, or ATM) on a blood-based or tissue-based assay
* History of bilateral orchiectomies or ongoing GnRH agonist or antagonist
* Castration-resistant disease based on progression per Prostate Cancer Working Group 2.21
* Prior treatment for metastatic prostate cancer with docetaxel and either abiraterone acetate or enzalutamide, OR ineligible for or declines treatment with docetaxel, abiraterone acetate, or enzalutamide.
* Adequate renal function with a serum creatinine ≤ 2.0 mg/dL or an estimated or calculated creatinine clearance of > 50 mL/min (calculated using the formula of Cockcroft and Gault)
* Adequate hepatic function with total bilirubin ≤ 1.5x the upper limit of normal (ULN) and ALT and AST less than 3x the ULN.
* Adequate hematological function with ANC ≥ 1500/mm3, hemoglobin ≥ 9.0 g/dL, and platelet count ≥ 100,000/mm3
* Age ≥ 18 years
* ECOG performance status of 0 or 1
* Ability to understand and the willingness to sign a written informed consent document
* Patients/participants with female partners of childbearing potential are eligible to participate if they agree to ONE of the following for the duration of the study:

  * Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent for duration of the study.
  * Agree to use a male condom and have their partner use a contraceptive method with a failure rate of <1% per year (intrauterine device or hormonal implant).
* Patients/participants must refrain from donating sperm for the duration of the study.
* Patients/participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile penetration for the duration of the study.

Exclusion Criteria:

* Participants who have received more than two prior chemotherapy regimens for metastatic castration-resistant prostate cancer.
* Participants who have any previous treatment with PARP inhibitors
* Participants who are receiving any other investigational agents.
* Participants who have received radiation therapy within 2 weeks or radionuclide treatment within 6 weeks prior to registration on this study
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to telaglenastat or talazoparib
* Concurrent use of moderate or strong CYP3A4 inducers or inhibitors, which could affect talazoparib plasma concentrations
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients known to be positive for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of objective responses | Measured from the start of the treatment through study completion, an average of 1 year
  Assessed by RECIST1.1
Rate of participants with clinical benefit | Measured from the start of the treatment through study completion, an average of 1 year
  Assessed by RECIST1.1
Rate of complete responses | Measured from the start of the treatment through study completion, an average of 1 year
  Assessed by RECIST1.1
Rate of partial responses | Measured from the start of the treatment through study completion, an average of 1 year
  Assessed by RECIST1.1
Rate of participants with progressive disease | Measured from the start of the treatment through study completion, an average of 1 year
  Assessed by RECIST1.1
Rate of participants with stable disease | Measured from the start of the treatment through study completion, an average of 1 year
  Assessed by RECIST1.1

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | 12 weeks
  The number and proportion of adverse events, graded as defined by CTCAE version 5.0 will be tabulated by type and grade. This analysis will be performed overall and separately for Cohort 1 and 2. Within a given patient, a given adverse event will be counted only once at the highest grade.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Lee, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation